CLINICAL TRIAL: NCT05613231
Title: Increasing Aerobic and Muscle-strengthening Physical Activity in Latinas Via Interactive Web-based Technology
Brief Title: Web-based Muscle-strengthening and Aerobic Physical Activity Intervention for Latinas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tanya Benitez, Assistant Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2104002972; R03CA252500 (NIH)
Record Dates: First submitted 2022-10-28; First posted 2022-11-14 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Inactivity, Physical
Keywords: physical activity; muscle-strengthening activity; strength training; Latinas; women; intervention; Internet
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic plus Muscle-Strengthening Activity Intervention (Experimental): Participants will receive access to a web-based, individually tailored, theory-driven aerobic moderate-to-vigorous physical activity (MVPA) intervention that was enhanced with content on muscle-strengthening activity.
  Interventions: Behavioral: Aerobic plus muscle-strengthening physical activity intervention
- Original Physical Activity Intervention (Active Comparator): Participants will receive access to a web-based, individually tailored, theory-driven aerobic moderate-to-vigorous physical activity (MVPA) intervention
  Interventions: Behavioral: Original physical activity intervention

INTERVENTIONS:
Behavioral: Aerobic plus muscle-strengthening physical activity intervention — The intervention is a 12-week Spanish language, Internet-based intervention promoting both aerobic and muscle-strengthening physical activity for Latina women.
  Arms: Aerobic plus Muscle-Strengthening Activity Intervention
Behavioral: Original physical activity intervention — The intervention is a 12-week Spanish language, Internet-based intervention promoting aerobic physical activity for Latina women.
  Arms: Original Physical Activity Intervention

SUMMARY:
The disproportionately low physical activity (PA) in Latinas, particularly muscle-strengthening activities, and related chronic diseases (e.g., obesity, diabetes, cancer) signifies an urgent public health concern. To address the lack of interventions promoting muscle-strengthening activities exclusively for Latinas, the investigators are testing the preliminary efficacy of a culturally and linguistically relevant, web-based aerobic plus muscle-strengthening PA intervention in this at-risk population. The web-based intervention provides a more comprehensive and highly disseminable approach for reducing PA-related health disparities in Latinas.

DETAILED DESCRIPTION:
Cancer is the leading cause of death among Latinos in the U.S. While engaging in a physically active lifestyle is one of the most important modifiable behaviors for reducing cancer risk; few Latinas achieve health-enhancing levels of physical activity (PA) recommended by the National PA Guidelines, particularly for muscle strengthening activities (MSA). For instance, 44% of Latinas meet the national guidelines for aerobic PA but only 17% meet the full guidelines for both aerobic and MSA. While the benefits of aerobic MVPA are well established for cancer and chronic disease prevention, participating in regular MSA may be key to further reducing cancer risk, as adherence to MSA guidelines has been associated with a 19% to 31% lower cancer mortality risk, independent of aerobic PA. There is a need for interventions promoting MSA in Latinas. However, only a select few MSA interventions have included Latinas in their sample, and none to the investigators' knowledge, were designed exclusively for this population or addressed socio-cultural factors influencing Latinas' muscle strengthening behaviors (e.g., perception that MSA is for men; MSA is an avoided topic in their culture and social circles; belief that women should only do certain types of MSA). Moreover, existing interventions often involved in-person exercise programs, which can be inaccessible to many Latinas due to barriers such as lack of transportation or fear of immigration enforcement. The research team has previously developed and tested aerobic moderate-to-vigorous PA (MVPA) interventions for Latinas that overcome barriers to in-person programs and address PA-related socio-cultural factors. These theory-driven, individually tailored interventions have shown success at increasing aerobic MVPA among Latina women in both print and Internet-based randomized controlled trials, and now provide an ideal platform for promoting MSA in this at-risk population. To address the gap in literature on MSA, the investigators recently conducted qualitative interviews with 19 Latinas to identify theory-based barriers and facilitators of muscle strengthening PA, then developed MSA intervention materials and further refined them for cultural appropriateness, relevance, and appeal in Latinas. In the proposed research, the investigators will incorporate the newly developed MSA promotion materials into the existing web-based aerobic MVPA intervention and conduct a 12-week fully online randomized pilot trial testing the preliminary efficacy of the newly adapted web-based aerobic plus MSA intervention for Latinas. Fifty Latina adults (i.e., aged 18-65 years) will be randomized to either the: 1) original aerobic MVPA intervention arm, or 2) aerobic MVPA plus MSA intervention arm. This study aims to: 1) Assess the preliminary efficacy of the aerobic plus MSA intervention for increasing MSA, and 2) Explore potential mediators and moderators of MSA. This interactive and highly disseminable approach can achieve significant health improvements in an at-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Sedentary (Less than 60 minutes per week of moderate or vigorous physical activity)
* Self-identify as Hispanic or Latino (or of a group defined as Hispanic/Latino by the Census Bureau
* Must be able to read and write Spanish fluently
* 18 - 65 years of age
* Have regular access to an Internet-connected device through home, work, or their community (e.g., public library, community center, neighbor's house) and video capabilities on cell phone, tablet, computer, for baseline and 12-week assessments.

Exclusion Criteria:

* Any orthopedic condition that would limit mobility
* History of heart disease, stroke or any other health condition that would make physical activity unsafe
* BMI above 45 kg/m2
* Current or planned pregnancy in the next 12 weeks
* Does not have regular access to an Internet-connected device

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Change in physical activity as reported by the 7-Day Physical Activity Recall (PAR) from baseline to week 12. | Baseline and week 12
  The 7-Day PAR is an interviewer administered instrument that uses multiple strategies for increasing accuracy of participant recall regarding many types of activities such as time spent sleeping and moderate, hard, and very hard intensity activities.
Change in muscle strengthening activities as reported by the Modifiable Physical Activity Questionnaire (MAQ) | Baseline and week 12
  The MAQ will assess frequency, intensity and duration of muscle strengthening activity

SECONDARY OUTCOMES:
Change in objectively measured physical activity as reported by ActiGraph accelerometer wear. | Baseline and week 12
  For the week prior to each assessment, participants will wear an Actigraph GT3X+ accelerometer which collects min/week of objectively measured MVPA
Change in upper body strength will be assessed by the one-minute repeated push-up test from baseline to week 12. | Baseline and week 12
  Participants will complete a 1-minute repeated push-up test via Zoom video that will be used as an objective measure upper body strength.
Change in lower body strength will be assessed by the one-minute repeated squat test from baseline to week 12.. | Baseline and week 12
  Participants will complete a 1-minute repeated squat test via Zoom video that will be used as an objective measure upper body strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University, Providence, Rhode Island, United States